CLINICAL TRIAL: NCT04303793
Title: Procedural Outcomes of Percutaneous PDA Closure: Comparative Study Between Different Devices.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Moheb El-Din, Assistant lecturer of cardiovascular medicine, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: congenital heart disease
Record Dates: First submitted 2020-03-07; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Percutaneous PDA closure — transcatheter patent ductus arteriosus closure

SUMMARY:
To compare safety, efficacy and procedural outcome of percutaneous PDA closure using different approaches for better characterization of device selection criteria.

ELIGIBILITY:
Inclusion Criteria:

* all patients who are candidate for transcatheter PDA closure

Exclusion Criteria:

1. Patients with PDA dependent pulmonary circulation.
2. Patients with small sized PDA which is silent by auscultation
3. Patients with large sized PDA which is unsuitable for Trans-catheter closure
4. Patients with PDA and severe irreversible pulmonary hypertension (Eisenmenger's syndrome) (7).
5. Patients with active infection or active infective endarteritis.
6. Patients refusing the study.

Ages: 1 Month to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Procedural safety | one month
  studying the occurrence of catheter related complications including
  1. Occurrence of vascular access hematoma(Yes/No )
  2. Occurrence of contrast induced nephropathy (Yes/No)
  3. PDA closure Device embolization (Yes/No)
  4. Cardiac tamponade (Yes/No)
Procedural efficacy | one month
  timing of complete closure of the PDA with no residual shunts
  1. Residual left to right shunt (Yes/No)
  2. Degree of the residual shunt (Trace, Mild , Moderate, severe)
  3. Timing of closure of the shunt( immediately postprocedural, 24 hours post procedural , 1 month post procedural )
Procedural outcomes | one month
  comparison of echocardiography data that will be done pre catheter closure, one day post procedure and one month later ( left ventricular and atrial dimensions-left ventricular ejection fraction-pulmonary artery systolic pressure- degree of tricuspid regurge)